CLINICAL TRIAL: NCT01568957
Title: Training Dual-Task Walking After Stroke: Effects on Attentional and Locomotor Control
Brief Title: Training Dual-Task Walking After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11SDG7270001
Record Dates: First submitted 2012-03-25; First posted 2012-04-02 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Stroke
Keywords: Gait; Dual-task; Obstacle avoidance; Attention allocation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dual-task gait training (Experimental): Gait training with simultaneous performance of cognitive tasks for 75% of training session.
  Interventions: Behavioral: Gait training
- Single-task gait training (Active Comparator): Gait training (without simultaneous cognitive task performance)
  Interventions: Behavioral: Gait training

INTERVENTIONS:
Behavioral: Gait training — Twelve 30-minute sessions plus 10-minute stretching and warm up, provided 3 times per weeks for 4 weeks. Up to 6 weeks are allowed to complete the 12 sessions.

SUMMARY:
Community ambulation is a highly complex skill requiring the ability to adapt to increased environmental complexity and perform multiple tasks simultaneously. Deficits in dual-tasking may severely compromise the ability to participate fully in community living. Unfortunately, current rehabilitation practice for stroke fails to adequately address dual-task limitations; individuals with stroke continue to exhibit clinically significant dual-task costs on gait at discharge. As a result, many stroke survivors are living in the community with residual deficits that may increase disability in the real world and lead to falls with devastating consequences. To address this issue, the proposed study investigates the efficacy of dual-task gait training on attention allocation and locomotor performance in community-dwelling stroke survivors. Because walking in the real world often requires time-critical tasks and obstacle avoidance, the investigators will test the impact of dual-task gait training on cognitive-motor interference during walking at preferred speed and at maximal speed (Aim 1), and on locomotor control during obstacle negotiation (Aim 2). The investigators will also evaluate the effects of the intervention on community reintegration and participation (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Within 3 years of stroke onset
* Living in the community, operationally defined as living in one's own home, or the home of a friend, relative, or caregiver
* Walking speed 0.6-1.1 m/s determined during 10-meter walk test
* Walk without the assistance of another person
* Medically stable and approved for participation by study physician
* Intact global cognition indicated by score > 23 on Montreal Cognitive Assessment
* Living in the community prior to stroke

Exclusion Criteria:

* Pre-existing neurological disorders (e.g., Parkinson's disease, Multiple Sclerosis, dementia, traumatic brain injury)
* Previous stroke with residual motor deficit
* Uncontrolled hypertension
* Inability to follow 3-step command
* Primary uncontrolled hearing impairment
* Severe uncontrolled visual impairment
* Any speech-language impairment affecting ability to respond verbally to auditory stimuli
* Timed Up and Go test > 15 seconds
* Lower extremity amputation
* Any orthopedic problem affecting gait
* Concurrent participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-09; Primary Completion 2017-03-29 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Dual-task cost on gait speed | 4 weeks
  The dual-task cost represents the difference between single and dual-task walking speed.

SECONDARY OUTCOMES:
Executive function | Measured at baseline, post intervention (4 weeks), 6 months post intervention
  A computerized version of the Stroop task will be used to assess changes in executive function.
Spontaneous physical activity | Measured at baseline, post intervention (4 weeks), 6 months post intervention
  Spontaneous physical activity will be assessed with an activity monitor (PAMSys) worn for two consecutive days at each assessment timepoint.
Kinematics of gait during obstacle crossing | Measured at baseline, post intervention (4 weeks), 6 months post intervention
Stroke Impact Scale | Measured at baseline, post intervention (4 weeks), 6 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Prudence Plummer, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Plummer-D'Amato P, Kyvelidou A, Sternad D, Najafi B, Villalobos RM, Zurakowski D. Training dual-task walking in community-dwelling adults within 1 year of stroke: a protocol for a single-blind randomized controlled trial. BMC Neurol. 2012 Oct 31;12:129. doi: 10.1186/1471-2377-12-129. PMID 23113928